CLINICAL TRIAL: NCT02224313
Title: Effect of Oral Estradiol and Progesterone Therapy on Vaginal Cytokines in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intira Sriprasert (Other)
Collaborators: TherapeuticsMD (Industry)
Responsible Party: Sponsor-Investigator, Intira Sriprasert, Dr., Eastern Virginia Medical School
Organization: Eastern Virginia Medical School (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRC-VgCy
Record Dates: First submitted 2014-07-30; First posted 2014-08-25 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Menopause
Keywords: vaginal cytokine
MeSH Terms: interventions — Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.Premenopausal women (No Intervention): No treatment
- 2.Postmenopausal women with hormones (Experimental): Oral hormone therapy will be given to women in this group. Daily dose of oral "estradiol" 1 mg will be given the first 14 days after enrollment. Then a daily dose of oral "estradiol" 1 mg and "progesterone" 100 mg for 14 days will be given during the following 14 days.
  Interventions: Drug: oral estradiol 1.0 mg; Drug: oral progesterone 100 mg

INTERVENTIONS:
Drug: oral estradiol 1.0 mg — one tablet of oral estradiol 1.0 mg once a day for 28 days
  Other Names: Estrace
  Arms: 2.Postmenopausal women with hormones
Drug: oral progesterone 100 mg — one tablet of oral progesterone 100 mg once a day for 14 days
  Other Names: Prometrium
  Arms: 2.Postmenopausal women with hormones

SUMMARY:
The purpose of this study is to compare the vaginal health between premenopausal and postmenopausal women before and after using oral "estradiol" for 14 days then "estradiol" and "progesterone" for 14 days.

DETAILED DESCRIPTION:
This research project recruits 10 healthy, premenopausal women (aged 20-40 years-old) with regular menstrual cycle with interval of 24-35 days and duration of 2-7 days and 10 healthy postmenopausal women (aged 45-60 years-old) with an intact uterus and at least 12 months but not more than 36 months of spontaneous amenorrhea.

Premenopausal women will not receive any study medication(s). Postmenopausal women will be assigned the intervention described below.

• Oral "estradiol" 1.0 mg tablet for 14 days, then oral "estradiol" 1.0 mg tablet and "progesterone" 100 mg capsule for 14 days

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal and Postmenopausal women:

  1. Female between the ages of 20 and 40 years (premenopausal arm), OR be a female between the ages of 45 and 65 years (postmenopausal arm) willing to participate in the study, as documented by signing the informed consent form.
  2. Postmenopausal women with an intact uterus and at least 12 months of spontaneous amenorrhea (postmenopausal arm), OR be a premenopausal women with regular menstrual cycle with interval of 24-35 days and duration of 2-7 days (premenopausal arm).
  3. No oral hormone therapy for 8 weeks and transdermal or vaginal hormone therapy for 4 week prior to the study.
  4. Willing to use oral hormone therapy during the study period (postmenopausal women only).
  5. Willing to abstain from using products (other than study medication) that contain estrogen, progestin, or progesterone throughout study participation.
  6. Have general good health.
  7. Willing to refrain from sexual intercourse for 48 hours before vaginal sample collection.
  8. Willing to abstain from use of vaginal product 7 days before vaginal sample collection.

Exclusion Criteria:

* To participate in the study, a subject must NOT

  1. Be allergic to estrogen or progesterone products
  2. Have active genital infection or inflammation based on vaginal wet preparation, power of hydrogen (pH), whiff test and potassium hydroxide (KOH) preparation 2.1 Vulvovaginal candidiasis, trichomonas vaginitis or bacterial vaginitis 2.2 Sexually transmitted diseases including herpes simplex viral infection, gonorrhea and Chlamydia
  3. Have a known contraindication for oral hormone therapy or allergy to use of estradiol and/or progesterone
  4. Have used estrogen alone or estrogen/progestin for any of the following time periods:

     4.1 Vaginal hormone products (ring, cream, gels) within 30 days prior to screening 4.2 Transdermal estrogen alone or estrogen/progestin products within 4 weeks prior to screening 4.3 Oral estrogen and/or progestin therapy within 8 weeks prior to screening 4.4 Progestational implants, estrogen or estrogen/progestational injectable drug therapy within 3 months prior to screening 4.5 Estrogen pellet therapy or progestational injectable drug therapy within 6 months prior to screening 4.6 Percutaneous estrogen lotions/gels within 4 weeks prior to screening
  5. Have used tamoxifen, raloxifene or other selective estrogen receptor modulators (SERMs) therapy within 8 weeks prior to screening
  6. Have used an intrauterine device (IUD) within 8 weeks prior to screening
  7. Have used vaginal products (pessary, tampon, tablets, douching) within 7 days prior to screening
  8. Have evidence of cervical, vaginal, or vulvar intraepithelial neoplasia or cancer
  9. Have a past or current history breast cancer, endometrial cancer or endometrial hyperplasia, hypertriglyceridemia or venous thromboembolism
  10. Be an immuno-compromised patient including those with human immunodeficiency viral infection, chronic glucocorticoid use or active treatment with immunosuppressive agents
  11. Have a history of or current evidence of thromboembolism
  12. Have evidence of uncontrolled Hypertension Blood pressure >140/100 mmHg
  13. Have confirmed Diabetes Mellitus
  14. Currently smoking
  15. For sexually active premenopausal women, should be protected against pregnancy by sterilization, condom use, abstinence, or same sex relationship

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Archer, MD, Study Director — Eastern Virginia Medical School
Locations (1):
- David Archer, MD, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.Premenopausal Women: Premenopausal women with no treatment assigned
Period: Overall Study
Arm/Group | 1.Premenopausal Women | 2.Postmenopausal Women With Hormones
Started | 10 | 10
Completed | 7 | 9
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Premenopausal Women: Premenopausal women at baseline
- Postmenopausal Women: Postmenopausal women at baseline
- Total: Total of all reporting groups
Arm/Group | Premenopausal Women | Postmenopausal Women | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.90 (5.11) | 56.44 (3.57) | 44.17 (4.34)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.06 (5.82) | 29.97 (6.71) | 30.02 (6.08)
Vaginal power of hydrogen (pH) [Mean (Standard Deviation); unit: pH] | 4.08 (0.17) | 6.33 (0.79) | 5.21 (0.48)

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Cytokines at Baseline
Description: Determine the differences in vaginal cytokines: interleukin (IL)-1β and IL-8 between premenopausal and postmenopausal women.
Time Frame: At baseline visit
Population: One postmenopausal women was excluded due to non-compliance of assigned intervention.
Measure: Mean (Standard Deviation); unit: pg/ug protein
Groups:
- Premenopausal Women: Premenopausal women in the study
- Postmenopausal Women: Postmenopausal women in the study
Arm/Group | Premenopausal Women | Postmenopausal Women
Number analyzed (Participants) | 10 | 9
pg/ug protein
  IL-8 | 2.73 (3.67) | 3.19 (3.38)
  IL-1β | 0.12 (0.24) | 0.04 (0.04)

2. Secondary Outcome: Vaginal Cytokines During Follow-up
Description: Determine the changes in vaginal cytokines in postmenopausal women following treatment with estradiol then estradiol and progesterone compared to the normal menstrual cycle changes in young premenopausal women.
Time Frame: At 14 days and 28 days follow-up
Population: Three premenopausal women were excluded due to missing data.
Measure: Mean (Standard Deviation); unit: pg/ug protein
Arm/Group | Premenopausal Women | Postmenopausal Women
Number analyzed (Participants) | 7 | 9
pg/ug protein
  IL-8 at 14 days | 0.92 (1.40) | 1.34 (0.96)
  IL-1B at 14 days | 0.02 (0.03) | 0.04 (0.07)
  IL-8 at 28 days | 0.69 (0.33) | 1.69 (1.70)
  IL-1B at 28 days | 0.04 (0.02) | 0.03 (0.04)

ADVERSE EVENTS:
Time Frame: We evaluated the adverse event at 14 days and 28 days follow-up visits.
Arm/Group | Premenopausal Women | Postmenopausal Women
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Several limitations of this study were the small sample size and limited follow-up time, which limited the power to detect statistical significance in some outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT02224313/Prot_SAP_000.pdf